CLINICAL TRIAL: NCT01572974
Title: Quality of Life in Barrett's Esophagus and GERD:GERD Symptoms, Perception of Cancer Risk, and Actual Cancer Risk
Brief Title: Quality of Life in Barrett's Esophagus and Gastro-Esophageal Reflux Disease
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: PS0056
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux Disease
Keywords: Barrett's esophagus; Gastroesophageal reflux disease; Quality of life
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No Barrett's esophagus: Subject without columnar lined esophagus
- Nondysplastic BE: Subject with columnar lined esophagus and absence of dysplasia
- Low grade dysplastic BE: subject with columnar lined esophagus and presence of low grade dysplasia
- High grade dysplastic BE: subject with columnar lined esophagus and presence of high grade dysplasia

SUMMARY:
To Compare the overall quality of life of patients with no Barrett's esophagus , non-dysplastic Barrett's Esophagus (NDBE), Barrett's esophagus with low grade dysplasia (LGD), and Barrett's esophagus with high grade dysplasia (HGD). We also Compare the overall quality of life of Barrett's esophagus patients with severe gastroesophageal reflux disease (GERD) symptoms to those with no GERD symptoms

DETAILED DESCRIPTION:
The presence of GERD symptoms is associated with a significant decrease in quality of life.While a diagnosis of Barrett's esophagus is also associated with a decrease in quality of life, these studies evaluated Barrett's esophagus patients with GERD symptoms.It is unclear whether decrements in quality of life from cancer risk in patients with Barrett's esophagus are due to actual cancer risk or a patient's false perception.Here we Compare the overall quality of life of patients with no Barrett's esophagus , non-dysplastic Barrett's Esophagus (NDBE), Barrett's esophagus with low grade dysplasia (LGD), and Barrett's esophagus with high grade dysplasia (HGD). The Investigators will also Compare the overall quality of life of Barrett's esophagus patients with severe gastroesophageal reflux disease (GERD) symptoms to those with no GERD symptoms. Finally the investigators will compare the overall quality of life of patients with a perceived low risk of esophageal cancer to those with a perceived high risk of esophageal cancer

ELIGIBILITY:
Inclusion Criteria:

Age 18 or above

At least one of the following:

Previous diagnosis of Barrett's esophagus Presence of GERD symptoms per patient report

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is a Veteran population presenting to a VA Hospital with GERD symptom or Barrett's esophagus
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2010-01; Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Health State Utility as measured by the Time Trade-off (TTO) method/Standard Gamble (SG) method | 1 year
  questionnaire

SECONDARY OUTCOMES:
SF-36 physical function (PF) subscale | 12 months
  questionnaire
SF-36 role limitations-physical (RP) subscale | 12 months
  questionnaire
SF-36 general health (GH) subscale | 12 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Medical Center
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Gerson LB, Ullah N, Hastie T, Triadafilopoulos G, Goldstein M. Patient-derived health state utilities for gastroesophageal reflux disease. Am J Gastroenterol. 2005 Mar;100(3):524-33. doi: 10.1111/j.1572-0241.2005.40588.x. PMID 15743346
- [Background] Crockett SD, Lippmann QK, Dellon ES, Shaheen NJ. Health-related quality of life in patients with Barrett's esophagus: a systematic review. Clin Gastroenterol Hepatol. 2009 Jun;7(6):613-23. doi: 10.1016/j.cgh.2009.02.024. Epub 2009 Mar 10. PMID 19281858
- [Background] Eloubeidi MA, Provenzale D. Health-related quality of life and severity of symptoms in patients with Barrett's esophagus and gastroesophageal reflux disease patients without Barrett's esophagus. Am J Gastroenterol. 2000 Aug;95(8):1881-7. doi: 10.1111/j.1572-0241.2000.02235.x. PMID 10950030
- [Background] Shaheen NJ, Green B, Medapalli RK, Mitchell KL, Wei JT, Schmitz SM, West LM, Brown A, Noble M, Sultan S, Provenzale D. The perception of cancer risk in patients with prevalent Barrett's esophagus enrolled in an endoscopic surveillance program. Gastroenterology. 2005 Aug;129(2):429-36. doi: 10.1016/j.gastro.2005.05.055. PMID 16083700
- [Background] Kruijshaar ME, Siersema PD, Janssens AC, Kerkhof M, Steyerberg EW, Essink-Bot ML; CYBAR Study Group. Patients with Barrett's esophagus perceive their risk of developing esophageal adenocarcinoma as low. Gastrointest Endosc. 2007 Jan;65(1):26-30. doi: 10.1016/j.gie.2006.05.030. PMID 17185076
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Kulig M, Leodolter A, Vieth M, Schulte E, Jaspersen D, Labenz J, Lind T, Meyer-Sabellek W, Malfertheiner P, Stolte M, Willich SN. Quality of life in relation to symptoms in patients with gastro-oesophageal reflux disease-- an analysis based on the ProGERD initiative. Aliment Pharmacol Ther. 2003 Oct 15;18(8):767-76. doi: 10.1046/j.1365-2036.2003.01770.x. PMID 14535869